CLINICAL TRIAL: NCT04652544
Title: Vitamin D Supplementation in Individuals With a Chronic Spinal Cord Injury - a Placebo-controlled Randomized Double-blinded Study
Brief Title: Vitamin D Supplementation in Individuals With a Chronic Spinal Cord Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-06
Record Dates: First submitted 2020-11-24; First posted 2020-12-03 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injuries; Vitamin D Deficiency
MeSH Terms: conditions — Spinal Cord Injuries; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Participants having a vitamin D status ≤ 75 nmol/L at baseline, will be randomly assigned to one of the three intervention groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Low" dose (Experimental): One vial with 600 µg cholecalciferol (corresponding to a total of 24'000 IU vitamin D) and one vial with placebo every month.
  Interventions: Drug: Cholecalciferol (Vitamin D3); Other: Placebo
- "High" dose (Experimental): Two vials with 600 µg cholecalciferol each (corresponding to a total of 48'000 IU vitamin D) every month.
  Interventions: Drug: Cholecalciferol (Vitamin D3)
- Placebo (Placebo Comparator): Two vials with a placebo every month.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cholecalciferol (Vitamin D3) — Vi-De 3® Monthly Dose from Dr. Wild & Co. AG (Muttenz, Switzerland) is a commercially available vitamin D3 supplement.
  Other Names: Vi-De 3® Monthly Dose
  Arms: "High" dose; "Low" dose
Other: Placebo — A placebo will be produced, consisting of the same ethanol solution as Vi-De 3® Monthly Dose, but without cholecalciferol.
  Arms: "Low" dose; Placebo

SUMMARY:
The main objective of this placebo-controlled randomized double-blinded study is to investigate the effect of vitamin D supplementation on vitamin D status (25(OH)D concentration in the blood) among individuals with a chronic spinal cord injury (SCI). Further, the effects of vitamin D supplementation on several other parameters (e.g. bone density and mood) are investigated, which could reveal positive secondary effects of supplementation that are especially relevant for clinical practice.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the influence of vitamin D supplementation among individuals with chronic SCI. The primary aim is to study whether different dosages (24'000 IU/month or 48'000 IU/month) of vitamin D supplementation over 12 months will lead to differences in vitamin D status as well as differences in several other outcomes. The use of a placebo group supports the evaluation of dose-response effects of vitamin D supplementation on the primary outcome (vitamin D status) and secondary outcomes (including bone density and mood) that are not only supported by randomized controlled trial standards but also informative in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent to the present study as documented by a signature
* Chronic (> 3 years) traumatic or non-traumatic spinal cord injury with a sub-C4-level lesion
* Wheelchair dependency during activities of daily living
* vitamin D status <75nmol/L

Exclusion Criteria:

* Contraindications to the investigational product
* Clinically relevant disorders,
* Pressure ulcer grade 3 or 4
* Pregnancy, breastfeeding
* Vitamin D supplementation (> 400 IU/day) within the last 12 months
* Visiting a country with increased sun exposure (below the 37th parallel north) within the last month before study enrolment or during the study
* Fractures in both arms and/or both legs within the last five years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Vitamin D status | 0 to 12 months
  Serum levels of 25(OH)D in nmol/L

SECONDARY OUTCOMES:
Bone density | At baseline and after 12 months
  Measurements of the forearm (radius), hip (femoral neck) and knee (distal femur and proximal tibia) will be performed using dual-energy X-ray absorptiometry (DXA) scans. T-values will be reported.
Mood | At 0, 3, 6, 9, 12 months
  Assessed by the Hospital Anxiety and Depression Scale (HADS) questionnaire, using a 4-step scale (1-4) with a total range of 14-56 and higher scores indicating worse outcomes.
Fatigue | At 0, 3, 6, 9, 12 months
  Assessed by the Fatigue Severity Scale (FSS) questionnaire, using a 8-step scale (1-7) with total range 9-63 and higher scores indicating worse outcomes.
Chronic pain | At 0, 3, 6, 9, 12 months
  The occurrence of pain since the last visit is assessed by one question of the SCI Secondary Conditions Scale (Kalpakjian, Scelza et al. 2007), providing a five-step rating (0-4) with a higher score indicating a worse outcome.
Recent pain | At 0, 3, 6, 9, 12 months
  The occurrence, kind, location and interference of pain during the last week is assessed using questions of the adapted version of the International SCI Pain Basic Data Set (Widerström-Noga, Biering-Sørensen et al. 2008). The interference of pain is measured on a 11-step scale (0-10), with total range 0-30 and higher scores indicating worse outcomes.
Pressure injuries | At 0, 3, 6, 9, 12 months
  The occurrence, localization and severity of pressure injuries is assessed by the exact questions of the first-wave questionnaire of the Swiss Spinal Cord Injury Cohort Study (SwiSCI) survey (Post, Brinkhof et al. 2011, Brinkhof, Fekete et al. 2016). The severity or grade is assessed using the European and US National Pressure Ulcer Advisory panels' (EPUAP-NPUAP) classification (National Pressure Ulcer Advisory Panel and Alliance. 2014), using a 4 point scale (1-4) and higher grades indicating worse outcomes.

OTHER OUTCOMES:
Handgrip strength | At 0, 3, 6, 9, 12 months
  The mean of three measurements of both hands will be measured in kg
Falls | At 0, 3, 6, 9, 12 months
  The incidence, reason (recreation or daily activity), possible injuries and care needed resulting from each fall since the last visit is assessed by several questions.
Functional independence | At 0, 3, 6, 9, 12 months
  Functional independence during daily living will be assessed by the Spinal Cord Independence Measure (SCIM, 3rd version)
Calcium status | At 0, 3, 6, 9, 12 months
  Serum levels of calcium (mmol/L) to monitor hypercalcemia
Parathyroid hormone status | At 0, 3, 6, 9, 12 months
  Serum levels of parathyroid hormone (ng/L) will be monitored as it is correlated to vitamin vitamin D status
Phosphate status | At 0, 3, 6, 9, 12 months
  Serum levels of phosphate (mmol/L) will be monitored as it is correlated to vitamin D status
Cystatin C status | At 0, 3, 6, 9, 12 months
  Serum levels of cystatin C (mg/L) to monitor kidney function
Estimated glomerular filtration rate (eGFR) status | At 0, 3, 6, 9, 12 months
  Serum levels of estimated glomerular filtration rate (eGFR) (mL/min) to monitor kidney function
Testosterone status | At 0, 3, 6, 9, 12 months
  Serum levels of testosterone (ng/dL) will be monitored as it is correlated to vitamin vitamin D status
Urinary tract infections | At 0, 3, 6, 9, 12 months
  The occurrence of urinary tract infections since the last visit is assessed by the exact questions of the first-wave questionnaire of the Swiss Spinal Cord Injury Cohort Study (SwiSCI) survey (Post, Brinkhof et al. 2011, Brinkhof, Fekete et al. 2016).
Sun exposure | At 0, 3, 6, 9, 12 months
  The time spent outdoors (min) with level of exposed skin during the last 7 days, following Hanwell et al (2010).
Skin phototype | At 0 months
  Six categories ranging from light to very dark skin types based on Fitzpatrick (1975)
SCI characteristics | At 0 months
  Time since SCI (years), neurological level of injury (NLI), and the degree of impairment following the American Spinal Injury Association (ASIA) Impairment Scale (AIS)
Personal characteristics | At 0, 3, 6, 9, 12 months
  Physical activity (hours and number of trainings), medication and nutritional supplements, and illnesses will be assessed by questionnaire. Weight will be measured on a scale.

CONTACTS AND LOCATIONS:
Overall Officials: Anke Scheel-Sailer, Dr. med., Principal Investigator — Head physician paraplegiology
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hertig-Godeschalk A, Flueck JL, Scheel-Sailer A, Perret C, Brinkhof MWG. No discernible effect of vitamin D supplementation on secondary outcomes in chronic spinal cord injury: Findings from a randomized controlled trial. J Spinal Cord Med. 2025 Oct 1:1-12. doi: 10.1080/10790268.2025.2557078. Online ahead of print. PMID 41032389
- [Derived] Hertig-Godeschalk A, Brinkhof MWG, Scheel-Sailer A, Perret C, Jenny A, Landmann G, Wyss PO, Flueck JL. Vitamin D supplementation in chronic spinal cord injury (VitD-SCI): study protocol for a randomised controlled trial. BMJ Open. 2021 Dec 17;11(12):e053951. doi: 10.1136/bmjopen-2021-053951. PMID 34921084